CLINICAL TRIAL: NCT05149027
Title: An Open-Label, Phase 1 Clinical Study to Evaluate the Safety, Tolerability, PK/PD and Preliminary Efficacy of HBM4003 in Combination With Toripalimab in Patients With Advanced HCC and Other Solid Tumors
Brief Title: A Study to Evaluate Safety, Tolerability, PK/PD and Preliminary Efficacy of HBM4003 Combine With Toripalimab in Patients With Advanced HCC and Other Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harbour BioMed (Guangzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4003.5
Record Dates: First submitted 2021-11-23; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBM4003+Toripalimap (Experimental): HBM4003 combined with toripalimab in patients with advanced HCC and other solid tumors
  Interventions: Drug: HBM4003 and Triprilimab

INTERVENTIONS:
Drug: HBM4003 and Triprilimab — Subjects will be treated with HBM4003 and Toripalimap on Day 1 during each 21-day cycles.

SUMMARY:
This is an open-label, multi-center phase 1 study. The trial, consisting of Part

1 dose confirmation and Part 2 dose expansion, is designed to evaluate the safety, tolerability, PK/PD and preliminary efficacy of HBM4003 in combination with Toripalimab in patients with advanced HCC and other solid tumors.

DETAILED DESCRIPTION:
subjects will be treated with HBM4003 in combination with Toripalimab for up to 2 years or until confirmed disease progression, unacceptable tolerability or treatment discontinuation through withdrawal of consent occurs, whichever happens first.

This trial consists of :

* A screening period: 28 days
* A treatment period:
* Part 1 dose confirmation study
* Part 2 dose expansion study
* A post-treatment follow-up period, including
* A safety follow-up period: 28 days after the last dose of study drug;
* Post-treatment follow-up visit: day 84 after the last dose of study drug;
* Survival follow-up.

ELIGIBILITY:
Main inclusion criteria :

1. Males or females aged ≥ 18 years at the time of signing the informed consent form. For Part 1 of this study, the subjects should be ≤ 75 years of age.
2. Patients for Part 1: patients histopathologically diagnosed with advanced or recurrent solid tumors or more line SOC failure or progression within 6m after adjuvant or neoadjuvant therapy.
3. For Part 2 of the study, patients with histopathologically confirmed advanced hepatocellular carcinoma; Barcelona Clinic Liver Cancer (BCLC) stage C or B; where stage B patients must be unsuitable for surgical and/or local therapy, or have progressive disease after surgical and/or local therapy, or refuse surgical and local therapy.

   1. Cohort 1: Patients with advanced HCC who have not received previous treatment with anti-PD-1 pathway drugs (including anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs), including patients who have received or have not received systemic treatment (e.g. anti-VEGF/VEGFR monoclonal antibodies, anti-VEGFR-TKIs, chemotherapy); patients who have received adjuvant/neoadjuvant therapy with anti-PD-1 pathway drugs and have disease progression more than 12 months after the end of treatment can be enrolled into this cohort
   2. Cohort 2: advanced HCC patients who have progressed during or after anti-PD-1 pathway drug therapy (with clearly documented radiographic evidence of progression), including patients who have or have not received systemic therapy (e.g., anti-VEGF/VEGFR monoclonal antibodies, anti-VEGFR-TKIs, chemotherapy); patients who have progressed within 6 months after the end of adjuvant/neoadjuvant therapy with anti-PD-1 pathway drugs may be enrolled into this cohort
   3. Other possible tumor expansion cohorts will be further revised as more data become available.
4. Patients must be able to provide fresh tumor tissues or archived tumor tissues.
5. Patients whose estimated survival time is more than 3 months.
6. Patients with at least one measurable lesion at baseline according to RECIST (Version 1.1).
7. Patients with Eastern Cooperative Oncology Group (ECOG) performance status score ≤ 1.
8. Patients whose organ function must meet the study requirements:
9. Every woman or man with potential fertility needs to use an effective contraceptive method.
10. Willing and able to comply with study-specified visits schedule, treatment plan, laboratory examination and other study procedures.

Main exclusion criteria:

1. Patients who are simultaneously participating in another clinical study, unless the study is an observational (non-interventional) clinical study or the patient is already in the survival follow-up period of the interventional study.
2. Patients with a history of severe allergic diseases, a history of severe drug allergies, and known or suspected allergy to macromolecular protein preparations or HBM4003 excipients or toripalimab excipients.
3. For the liver cancer cohort in Part 2 of the study, patients with pathological findings suggestive of fibrolamellar hepatocellular carcinoma, sarcomatoid hepatocellular carcinoma, cholangiocarcinoma, or mixed hepatocellular carcinoma-cholangiocarcinoma were excluded.
4. Previous and concomitant drugs or treatments to be excluded like CTLA4, PD-1,PD-L1.
5. Insufficient recovery from previous treatments
6. Diseases that may affect the efficacy and safety of the investigational product.
7. A history of other malignant diseases within 5 years before the first dose.
8. Symptomatic, active, or urgent treatment-requiring central nervous system (CNS) metastasis with imaging evidence (based on CT or MRI assessment).
9. Subjects with pleural effusion, pericardial effusion, or ascites
10. Patients with severe liver cirrhosis, liver atrophy or hypertension.
11. Imaging revealed that the main portal vein tumor thrombus was more than 1/2, and the vein tumor thrombus or heart was involved.
12. Grade ≥ 2 hepatic encephalopathy within 12 months, or currently requiring medication to prevent or control hepatic encephalopathy.
13. Patients who the investigator believes may have other factors that will affect the efficacy or safety evaluation of this study (e.g., mental disorders, alcoholism, drug use, etc.).
14. Women who are pregnant or breastfeeding, or who plan to become pregnant during the study period and within 3 months after the last administration of the investigational product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Part1:Number of subjects with DLT in each dose group within 1 cycles (21 days) after the first drug administration | approximate 21 days
  Number of subjects who experience DLT events
Part1:The maximum tolerated dose (MTD) of HBM4003 combined with toripalimab | approximate 21 days
Part1:Recommended Phase 2 dose (RP2D) of HBM4003 combined with toripalimab | approximate 21 days
Part2:ORR, as determined by the Investigator using RECIST 1.1 | maximum 2 years
  Proportion of subjects with complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Part 1:ORR, as determined by the Investigator using RECIST 1.1 for solid tumors, using RECIST 1.1 and mRECIST for HCC | maximum 2 years]
  Proportion of patients with complete response (CR) and partial response (PR)
Part 1: Disease Control Rate, DCR, as determined by the Investigator using RECIST 1.1 for solid tumors, using RECIST 1.1 and mRECIST for HCC | maximum 2 years
  including proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD)
Part 1: Duration of Response, DOR, as determined by the Investigator using RECIST 1.1 for solid tumors, using RECIST 1.1 and mRECIST for HCC | maximum 2 years
  Calculate the duration from the first confirmed CR or PR to the date of disease progression or death (for any reason)
Part 1: Duration of Disease Control, DDC, as determined by the Investigator using RECIST 1.1 for solid tumors, using RECIST 1.1 and mRECIST for HCC | maximum 2 years
  For subjects with Cr, PR or SD, the duration from the time of initial administration to the date of disease progression or death (for any reason) was calculated
Part2: ORR, as determined by the Investigator using mRECIST for HCC | maximum 2 years
  Proportion of patients with complete response (CR) and partial response (PR)
Part 2: Disease Control Rate, DCR, as determined by the Investigator using RECIST 1.1 and mRECIST for HCC | maximum 2 years
  including proportion of subjects with complete response (CR) and partial response (PR) and stable disease (SD)
Part2: Duration of Response, DOR, as determined by the Investigator using RECIST 1.1 and mRECIST for HCC | maximum 2 years
  Calculate the duration from the first confirmed CR or PR to the date of disease progression or death (for any reason)
Part2:Duration of Disease Control, DDC, as determined by the Investigator using RECIST 1.1 and mRECIST for HCC | maximum 2 years
  For subjects with Cr, PR or SD, the duration from the time of initial administration to the date of disease progression or death (for any reason) was calculated
Cmax | maximum 2 years
  Peak Plasma Concentration
Tmax | maximum 2 years
  Time to reach maximum serum concentration
AUC0-last | maximum 2 years
  Area under the plasma concentration versus time curve from time zero to last
AUC0-tau | maximum 2 years
  Area under the serum concentration versus time curve from time zero to the dosing interval tau
The immunogenicity of HBM4003 and Triprilimab | maximum 2 years
  Including the incidence of ADA positive. For ADA positive patients, the incidence of neutralizing antibody (NAB) was analyzed.
Part 2: Overall survival (OS) | maximum 2 years
  the length of time from the start of treatment to the death of the subject (for any reason)
Part 2: Progression-free survival (PFS) | maximum 2 years
  the length of time from the beginning of treatment to the beginning of disease progression or death (for any reason)

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Hao, Doctor, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital